CLINICAL TRIAL: NCT05907278
Title: The Advanced Cooking Education (ACE) 4-H After School Club: A Feasibility Study
Brief Title: Advanced Cooking Education Feasibility Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cornell University (Other)
Collaborators: United States Department of Agriculture (USDA) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 0009007
Record Dates: First submitted 2023-06-08; First posted 2023-06-18 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2023-06

CONDITIONS: Adolescent Behavior; Nutrition, Healthy
Keywords: Adolescents; Nutrition intervention; Culinary program
MeSH Terms: conditions — Adolescent Behavior

STUDY DESIGN:
Intervention Model Description: All participants receive the intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): The ACE Program is a culturally inclusive, 4-H after school club where youth meet once a week for 12 weeks virtually. They also receive groceries to make a meal 1 day a week.
  Interventions: Behavioral: Advanced Cooking Education

INTERVENTIONS:
Behavioral: Advanced Cooking Education — Participants attend the ACE Program for 12 weeks after school.
  On one assigned day of the week, participants attend ACE virtually. The session will begin with mindfulness exercises (15 minutes), professional development session (50 minutes), nutrition education lesson (20 minutes), and reflection period to talk about their experience in cooking lessons (25 minutes).
  On any day during the week, the students will make a dish using groceries they received (1 hour).

SUMMARY:
The aim of this study is to look at outcomes related to diet and nutrition, mindfulness, and cooking skills amongst middle school students who participated in a 12-week 4-H after school program called the Advanced Cooking Education Program.

DETAILED DESCRIPTION:
Participants are all assigned to the Advanced Cooking Education Program. Data collection was done before and after the program. The investigators hypothesize that after the program, adolescents' diet quality, cooking-related skills, stress levels will be improved compared to prior of the program.

ELIGIBILITY:
Inclusion Criteria:

* 7th and 8th grade students attending Title I funded schools in New York City
* Caregivers of 7th and 8th grade students attending Title I funded schools in New York City

Exclusion Criteria:

* Do not speak/understand English

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2021-09-13 (Actual); Primary Completion 2022-05-19 (Actual); Study Completion 2022-05-26 (Actual)

PRIMARY OUTCOMES:
Change in diet quality, measured by the Healthy Eating Index Scores | Baseline, 12 weeks [endpoint]
  Scores are calculated from three 24-hour diet records, range from 0-100. Higher score reflects higher alignment between one's diet and recommendations from Dietary Guidelines for Americans

SECONDARY OUTCOMES:
Change in body mass index | Baseline, 12 weeks [endpoint]
  Height will be measured using stadiometer to nearest decimal point in cm. Weight measured using scale to nearest decimal in kg. Body mass index calculated using kg/m^2.
Change in body fat percentage | Baseline, 12 weeks [endpoint]
  Measured using a scale to nearest decimal
Change in waist circumference | Baseline, 12 weeks [endpoint]
  Measured using a waist circumference tape to the nearest decimal in cm.
Change in dermal carotenoids level | Baseline, 12 weeks [endpoint]
  Measured using the Veggie Meter device, range from 0-800. Higher score acts as proxy for increased fruits and vegetables consumption.
Change in household food security | Baseline, 12 weeks [endpoint]
  Short form food security survey module by the USDA
Change in child food security | Baseline, 12 weeks [endpoint]
  Child version of food security survey module by the USDA
Change in culinary skills | Baseline, 12 weeks [endpoint]
  iCook program youth culinary skill survey with 5-point likert scale questions with higher scores indicate higher skill level (better outcome). Min=7, Max=35
Change in culinary attitudes | Baseline, 12 weeks [endpoint]
  Cooking with kids survey with 5-point likert scale questions with higher scores indicate more positive attitude (better outcome). Min=6, Max=30
Change in culinary self-efficacy | Baseline, 12 weeks [endpoint]
  iCook program youth culinary self-efficacy survey with 5-point likert scale questions with higher scores indicate higher self-efficacy (better outcome). Min=6, Max=30.
Change in perceived stress | Baseline, 12 weeks [endpoint]
  Used the Cohen perceived stress scale. Higher scores mean increased stress (worse outcome). Min=0, Max=40
Change in food neophobia | Baseline, 12 weeks [endpoint]
  FNTT10 survey with 5-point likert scale questions, higher scores mean less neophobia (better outcome). Min=10, Max=50.
Change in sense of purpose | Baseline, 12 weeks [endpoint]
  Used the Clarement Purpose Scale survey questions, higher scores mean higher sense of purpose (better outcome). Min=12, Max=60
Change in social and emotional competency | Baseline, 12 weeks [endpoint]
  Used the SEC survey by CASEL, higher scores mean higher competence (better outcome). Min=17, Max= 68
Change in family mealtime beliefs | Baseline, 12 weeks [endpoint]
  Calculated based on the Fulkerson family mealtime survey. A total of 9 questions that are scored independently. Each: Min=1, Max=4. Higher scores indicate better family mealtime practices (better outcome).

CONTACTS AND LOCATIONS:
Overall Officials: Tashara M Leak, PhD RD, Principal Investigator — Cornell University
Locations (1):
- Cornell University, Ithaca, New York, United States

IPD SHARING:
Plan to Share IPD: No